CLINICAL TRIAL: NCT01754597
Title: Evolution Natriuretic Peptide Concentrations of B-type (BNP) During General Anesthesia Under Propofol and Sevoflurane Association in Patients Previously Sensitized to Anthracyclines. Pilot Study in Patients Operated on for Breast Cancer.
Brief Title: Natriuretic Peptide Concentrations of B-type (BNP) During Anesthesia in Patients Previously Sensitized to Anthracyclines
Acronym: PEP-NAT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB2009-39
Record Dates: First submitted 2012-11-06; First posted 2012-12-21 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Anesthesia
MeSH Terms: conditions — Breast Neoplasms | interventions — pro-brain natriuretic peptide (1-76)

STUDY DESIGN:
Intervention Model Description: This feasibility study will describe the evolution of NT-ProBNP during general anesthesia in patients undergoing surgery for breast cancer, depending on whether or not they have previously been treated with anthracyclines.
  The data collected in this study will be used later in a clinical trial comparing the occurrence of subclinical heart failure during breast cancer surgery under general anesthesia, depending on whether patients have been sensitized to anthracyclines.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants not previously treated with anthracyclines (Other): No anthracycline treatment in the 6 months prior to inclusion.
  Interventions: Other: Dosage of B-type natriuretic peptide (NT-proBNP)
- Participants previously treated with anthracyclines (Other)
  Interventions: Other: Dosage of B-type natriuretic peptide (NT-proBNP)

INTERVENTIONS:
Other: Dosage of B-type natriuretic peptide (NT-proBNP) — NT-proBNP concentration assessed at the following time points :
  * T0: before induction of general anesthesia, NT-proBNP measurement
  * T1: 30 minutes after induction of general anesthesia
  * T2: at the end of the procedure
  * T3: in the postoperative period, 6 hours after the end of the procedure
  * T4: in the postoperative period, 24 hours after the end of the procedure

SUMMARY:
The cardiotoxicity of anthracyclines chemotherapy remains a major problem, despite clinical and echocardiographic monitoring. In the case of treatment for breast cancer, surgery requiring general anesthesia may follow chemotherapy. Although a possible interaction between general anesthetics and anthracyclines on systolic function is only rarely mentioned, some cases of heart failure and / or conduction disturbances peranesthésique were observed in patients treated or previously treated with anthracyclines. The determination of concentration of BNP is a diagnostic tool used in the detection of heart failure and acute coronary syndromes. The question of a possible synergism between cardiotoxic anthracyclines and anesthetic agents arises. Given its minimally invasive nature and its diagnostic value, the BNP assay might thus allow to highlight a possible subclinical deficiency. To our knowledge, there is very little data regarding a possible synergism between cardiotoxic anthracyclines and anesthetic agents.

DETAILED DESCRIPTION:
The cardiotoxicity of anthracyclines chemotherapy remains a major problem, despite clinical and echocardiographic monitoring. In the case of treatment for breast cancer, surgery requiring general anesthesia may follow chemotherapy. Although a possible interaction between general anesthetics and anthracyclines on systolic function is only rarely mentioned, some cases of heart failure and / or conduction disturbances peranesthésique were observed in patients treated or previously treated with anthracyclines. The determination of concentration of BNP is a diagnostic tool used in the detection of heart failure and acute coronary syndromes. In fact, it is one of the most sensitive markers of impaired myocardial function, and an increase in interest rates may precede any other biological changes. In a patient who received anthracycline, although it remains asymptomatic elevation of NT-proBNP concentration may persist for some months after exposure, and that, whatever the doses received. The question of a possible synergism between cardiotoxic anthracyclines and anesthetic agents arises. Given its minimally invasive nature and its diagnostic value, the BNP assay might thus allow to highlight a possible subclinical deficiency. To our knowledge, there is very little data regarding a possible synergism between cardiotoxic anthracyclines and anesthetic agents.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years with effective contraceptive method (if applicable)
* NT-proBNP <125 pg / ml
* ASA 1 or 2,
* Breast cancer histologically proven
* Mastectomy or lumpectomy
* Neoadjuvant chemotherapy with anthracyclines in 6 months or received no chemotherapy with anthracyclines,
* Patients who received the briefing and signed the informed consent
* Patients affiliated to a social security system.

Exclusion Criteria:

* Patients for whom the maintenance of general anesthesia does not use halogenated.
* Renal impairment: Creatinine clearance <60 ml / min,
* Patients who for reasons psychological, social, family or geographical could not be treated or monitored regularly according to the criteria of the study, patients deprived of liberty or under guardianship.
* Presence of a cardiopathy
* Pregnant Women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GEKIERE Jean Pierre, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Not Previously Treated With Anthracyclines: No anthracycline treatment in the 6 months prior to inclusion.
  Dosage of B-type natriuretic peptide (NT-proBNP): NT-proBNP concentration assessed at the following time points :
  * T0: before induction of general anesthesia, NT-proBNP measurement
  * T1: 30 minutes after induction of general anesthesia
  * T2: at the end of the procedure
  * T3: in the postoperative period, 6 hours after the end of the procedure
  * T4: in the postoperative period, 24 hours after the end of the procedure
Period: Overall Study
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines
Started | 29 | 25
Completed | 23 | 20
Not Completed | 6 | 5
Not completed — Dosage of NT-proBNP not performed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.4) | 49.3 (8.5) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Pre-operative Concentration of NT-proBNP
Description: Mean concentration of NT-proBNP measured before surgery.
Time Frame: Before breast surgery
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines
Number analyzed (Participants) | 23 | 20
pg/ml | 38.9 (27.0) | 32.2 (18.4)
Statistical Analysis 1: Comparison: Participants Not Previously Treated With Anthracyclines vs Participants Previously Treated With Anthracyclines; Test type: Superiority; p = 0.714, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Concentration of NT-proBNP at the End of Intervention
Description: Mean concentration of NT-proBNP measured at the end of intervention
Time Frame: At the end of breast surgery
Population: Participants with dosage available
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines
Number analyzed (Participants) | 22 | 20
pg/ml | 42.2 (28.0) | 34.6 (20.0)
Statistical Analysis 1: Comparison: Participants Not Previously Treated With Anthracyclines vs Participants Previously Treated With Anthracyclines; Test type: Superiority; p = 0.492, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Post-operative Concentration of NT-proBNP
Description: Mean concentration of NT-proBNP measured 24 hours after breast surgery
Time Frame: 24 hours after breast surgery
Population: Participants with NT-proBNP dosage available
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines
Number analyzed (Participants) | 23 | 20
pg/ml | 107.6 (79.1) | 75.9 (61.1)
Statistical Analysis 1: Comparison: Participants Not Previously Treated With Anthracyclines vs Participants Previously Treated With Anthracyclines; Test type: Superiority; p = 0.183, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24 hours after surgery
Description: Only mortality and serious adverse events were collected. These were collected in all included participants (29 +25 = 54 were included), and not only for those who completed the study (23 +20 = 43 completed the study) Non-serious adverse events were not collected.
Arm/Group | Participants Not Previously Treated With Anthracyclines | Participants Previously Treated With Anthracyclines
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes